CLINICAL TRIAL: NCT04385550
Title: A Randomized, Open-label, Controlled, Multicenter Phase III Study of Hydrochloride Capsule Combined With AK105 Injection Versus Standard Second-line Chemotherapy for Advanced Gastric and Gastro-oesophageal Junction Adenocarcinoma
Brief Title: A Study of Anlotinib Hydrochloride Capsule Combined With AK105 Injection in Subject With Advanced Gastric and Gastro-oesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AK05-III-01
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric and Gastro-oesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib hydrochloride capsule + AK105 injection (Experimental): Anlotinib hydrochloride capsule 12mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) plus AK105 200mg intravenously (IV) on Day 1 of each 21-day cycle.
  Interventions: Drug: Anlotinib hydrochloride capsule; Drug: AK105 injection
- Standard Second-line Chemotherapy (Active Comparator): Participants receive 80 mg/m² IV paclitaxel on Days 1, 8 and 15 of each 28-day cycle, or 75mg/m² docetaxel every 3 weeks of each 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel injection; Drug: Docetaxel injection

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsule — Anlotinib hydrochloride capsule 12mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Arms: Anlotinib hydrochloride capsule + AK105 injection
Drug: AK105 injection — AK105 200mg intravenously (IV) on Day 1 of each 21-day cycle.
  Arms: Anlotinib hydrochloride capsule + AK105 injection
Drug: Paclitaxel injection — Paclitaxel injection 80mg / m² IV on Days 1, 8 and 15 of each 28-day cycle.
  Arms: Standard Second-line Chemotherapy
Drug: Docetaxel injection — Docetaxel injection 75mg / m² IV every 3 weeks of each 21-day cycle.
  Arms: Standard Second-line Chemotherapy

SUMMARY:
This is a randomized, controlled, open-label, multicenter study to evaluate efficacy of AK105 injection combined with Anlotinib Hydrochloride Capsules versus standard second-line chemotherapy. Patients are treated with AK105 injection combined with Anlotinib Hydrochloride Capsules or standard second-line chemotherapy, with 1:1 random ratio.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understood and signed an informed consent form; 2.Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months; 3. Histopathology or cytology confirmed as metastatic or local advanced gastric and gastro-oesophageal junction adenocarcinoma; 4. First-line standard chemotherapy regimen in patients with advanced gastric or gastroesophageal junction adenocarcinoma after treatment failure; 5. Has at least one measurable lesion; 6. Weight ≥40 kg or BMI ≥18.5; 7. Adequate organ function; 8. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ;No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

Exclusion Criteria:

* 1. Histopathology confirmed as squamous cell carcinoma, carcinoid, undifferentiated carcinoma, or other gastric cancer; 2. HER2 positive; 3. Has received paclitaxel or docetaxel in the first-line treatment; 4. Has received paclitaxel or docetaxel in the neoadjuvant or adjuvant treatment regimen and have relapsed or metastasized within 6 months after the last dose; 5. Has other malignant tumors within 5 years; 6. Has used anti-angiogenic drugs such as anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, bevacizumab, or related immunotherapy drugs for PD-1, PD-L1, etc; 7. Severe hypersensitivity after administration of other monoclonal antibodies; 8. Has spinal cord compression, cancerous meningitis and symptomatic brain metastasis； 9. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1; 10. Has received radiotherapy, chemotherapy and surgery within 4 weeks before the first dose; 11. Has gastrointestinal bleeding tendency within 4 weeks before the first dose; 12. The tumor has invaded important blood vessels and will cause fatal bleeding; 13. Has multiple factors affecting oral medication; 14. Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage; 15. Has any active autoimmune disease or history of autoimmune disease; 16. Immunosuppressant or systemic or absorbable local hormone therapy is required to achieve the aim of immunosuppression (dose > 10mg/ day prednisone or other therapeutic hormones) and is still used within 2 weeks after the first administration; 17. Has any serious and / or uncontrolled disease; 18. Has active viral infection; 19. Has participated in other anticancer drug clinical trials within 4 weeks; 20. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 45 weeks
  OS defined as the time from randomization to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 45 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall response rate (ORR) | up to 45 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Disease control rate (DCR) | up to 45 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of response (DOR) | up to 45 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Shijitan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - The Sixth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Quanzhou First Hospital, Quanzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital,Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Cancer Hospital, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Hospital of Jiangnan University, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancar Hospital, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjing, Tianjing
  - Tianjin Medical University Cancer Institute and Hospital, Tianjing, Tianjing
  - The First People's Hospital of kashi region, Kashgar, XinJiang Uighur Autonomous Region